CLINICAL TRIAL: NCT02564913
Title: Integrated Clinical Evaluation of Traditional Chinese Medicine (TCM) and Conventional Medicine on Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Po-Chi Hsu, traditional Chinese medical doctor, Changhua Christian Hospital
Other Study IDs: 111106
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes Mellitus
Keywords: tongue diagnosis; heart rate variability; nailfold videocapillaroscopy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- control group
  Interventions: Other: clinical evaluation
- pre-DM group
  Interventions: Other: clinical evaluation
- DM group

INTERVENTIONS:
Other: clinical evaluation
  Groups: control group; pre-DM group

SUMMARY:
In traditional Chinese medicine (TCM), examination of the tongue plays an important role in diagnosis. The characteristics of the tongue(e.g., color of the tongue body, tongue fur, teeth-marked tongue) provides some clues and prognosis, which are considered a reflection of the body's internal condition. Diabetes mellitus is a metabolic disorder of hyperglycemia, which lead to damage the kidneys, eyes, nerves, blood vessels, and heart. Long standing hyperglycemia can also be associated with buccal alteration. The purpose of this study was to survey on tongue diagnosis and other examinations associated with diabetic mellitus.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients(ac sugar>126mg/dl or HbA1c>6.5, twice)
* pre-diabetic patients(100mg/dl <ac sugar<126mg/dl, or 5.9<HbA1c<6.5)
* non-diabetic patients(ac sugar<100mg/dl )

Exclusion Criteria:

* acute infectious disease,
* cancer,
* End Stage Renal Disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators recruited the control group , the pre-DM group, and the DM group.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2011-12; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
tongue diagnosis | 1 year
heart rate variability | 1 year
nailfold videocapillaroscopy | 1 year